CLINICAL TRIAL: NCT00566553
Title: The Effect of Grape Seed Extract on Estrogen Levels of Postmenopausal Women: A Pilot Study
Brief Title: The Effect of Grape Seed Extract on Estrogen Levels of Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dietlind Wahner-Roedler, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-009628
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: Grape Seed Extract; Breast Cancer; Estrogen Levels; Aromatase Inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Grape Seed Extract; Activins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Grape Seed Extract # 1 (Active Comparator): 200 mg [1 pill]
  Interventions: Dietary Supplement: Grape Seed Extract
- Grape Seed Extract # 2 (Active Comparator): 200 mg [2 pills]
  Interventions: Dietary Supplement: Grape Seed Extract
- Grape Seed Extract # 3 (Active Comparator): 200 mg [3 pills]
  Interventions: Dietary Supplement: Grape Seed Extract
- Grape Seed Extract # 4 (Active Comparator): 200 mg [4 pills]
  Interventions: Dietary Supplement: Grape Seed Extract

INTERVENTIONS:
Dietary Supplement: Grape Seed Extract — 200 mg dose daily for 12 weeks.
  Other Names: ActiVin®
  Arms: Grape Seed Extract # 1
Dietary Supplement: Grape Seed Extract — 400 mg dose daily for 12 weeks.
  Other Names: ActiVin®
  Arms: Grape Seed Extract # 2
Dietary Supplement: Grape Seed Extract — 600 mg dose daily for 12 weeks.
  Other Names: ActiVin®
  Arms: Grape Seed Extract # 3
Dietary Supplement: Grape Seed Extract — 800 mg dose daily for 12 weeks.
  Other Names: ActiVin®
  Arms: Grape Seed Extract # 4

SUMMARY:
The role of estrogens in the pathogenesis of breast cancer has been well documented. This has led to the development of "Anti-Estrogens" (selective estrogens receptor modulators and Aromatase Inhibitors), used for treatment and prevention of breast cancer. These agents, however, have significant side effects, which are not acceptable to many healthy high-risk women. There is preliminary evidence that grape seed extract acts as "natural" aromatase inhibitor (1). This study has the potential to quantify the effectiveness of a natural substance that mimics the action of pharmaceutical aromatase inhibitors.

DETAILED DESCRIPTION:
Early detection of breast cancer with screening mammography and the use of more effective medical therapies have led to a decrease in breast cancer mortality. However, breast cancer is still the second leading cause of cancer death in women (2). Therefore, the future lies in not only early detection but prevention of breast cancer. Currently available chemopreventive agents are associated with potentially serious side effects and can be quite costly, especially when taken for extended periods of time. Therefore, they are usually targeted only to women at high risk of disease. Identification of an inexpensive, efficacious preventive therapy with few or no side effects would represent a major advance in reducing the morbidity and mortality due to breast cancer. One exciting possibility is grape seed extract. Grapes and grape seeds contain procyanidins, a highly active subclass of flavonoids with actions similar to pharmaceutical aromatase inhibitors (AIs). These procyanidin dimers have been found to suppress estrogen biosynthesis both in vitro and in animal models (1). Based upon this knowledge we proposed this dose finding pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 - 75 years
* Able to understand and sign a consent form
* Postmenopausal (no menstrual period for 1 year or more)
* No personal cancer history (except for non-melanoma skin cancer)
* No hormone replacement therapy or anti-estrogens within 6 months of baseline

Exclusion Criteria:

* Known allergy to grapes or grape products
* Currently on ACE inhibitors, methotrexate, allopurinol, coumadin (Warfarin, Jantoven), heparin, clopidogrel (Plavix), or cholesterol lowering medication

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-02; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To document that grape seed extract taken orally will decrease plasma estrogen levels (estrone (E1), estradiol (E2), and E1-conjugates) and increase precursor androgen levels (testosterone and androstenedione) in healthy postmenopausal women. | 12 weeks

SECONDARY OUTCOMES:
To determine the most effective, well tolerated dose of grape seed extract resulting in a decrease in plasma estrogen levels (E1, E2, E1-conjugates) and increase in precursor androgens (testosterone and androstenedione). | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dietlind L. Wahner-Roedler, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Eng ET, Ye J, Williams D, Phung S, Moore RE, Young MK, Gruntmanis U, Braunstein G, Chen S. Suppression of estrogen biosynthesis by procyanidin dimers in red wine and grape seeds. Cancer Res. 2003 Dec 1;63(23):8516-22. PMID 14679019
- [Background] American Cancer Society. Cancer Facts and Figures 2005. Atlanta, GA: American Cancer Society; 2005.
- See also: American Cancer Society. Cancer Facts & Figures 2005. — http://www.cancer.org/acs/groups/content/@nho/documents/document/caff2005f4pwsecuredpdf.pdf